CLINICAL TRIAL: NCT01765959
Title: "Auricular Acupuncture and Cognitive Behavioral Therapy in the Context of Insomnia and Low Dose Dependence of Benzodiazepine-like Drugs and Other Sleep Medicine With Addiction Risk"
Brief Title: Auricular Acupuncture and Cognitive Behavioral Therapy Treatment for Insomnia
Acronym: NADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA2011-59
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Insomnia; Quality of Life
Keywords: Insomnia; Auricular acupuncture; CBT
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture, Ear; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular acupuncture (AA) (Active Comparator): Auricular acupuncture (AA) group will receive treatment twice a week for four weeks. Each session will take approximately 60 minutes in which there will be active treatment time for 40 minutes. During treatment the respondents will have 5 thin sterile, disposable steel needles superficially placed in each outer ear. Before needle insertion the outer ears will be cleaned with disinfection solution. During treatment the respondents will sit down in silence; with eyes shut and focus on a normal calm breathing. The acupuncturist will not be in the room during treatment. After 40 minutes the respondents remove the needles and put them in a box suited for disposed needles. If needed, assistance to remove needles will be given from the acupuncturist.
  Interventions: Other: Auricular acupuncture (AA)
- Cognitive behavioral therapy (CBT) (Active Comparator): Cognitive behavioral therapy (CBT) group will receive manual based sessions for sleeping disorders. The group meets once a week during six weeks according to following program:
  Session 1 - introduction, self-help concept Session 2 - biology of sleep, sleep restriction, Session 3 - stimulus control Session 4 - visualization as relaxation, Session 5 - how to deal with negative and automatic thoughts, Session 6 How to solve problems, planning for the future
  Interventions: Other: cognitive behavioral therapy (CBT)

INTERVENTIONS:
Other: Auricular acupuncture (AA) — Auricular acupuncture (AA) group will receive treatment twice a week for four weeks. Each session will take approximately 60 minutes in which there will be active treatment time for 40 minutes. During treatment the respondents will have 5 thin sterile, disposable steel needles superficially placed in each outer ear. Before needle insertion the outer ears will be cleaned with disinfection solution. During treatment the respondents will sit down in silence; with eyes shut and focus on a normal calm breathing. The acupuncturist will not be in the room during treatment. After 40 minutes the respondents remove the needles and put them in a box suited for disposed needles. If needed, assistance to remove needles will be given from the acupuncturist.
  Arms: Auricular acupuncture (AA)
Other: cognitive behavioral therapy (CBT) — Cognitive behavioral therapy (CBT) group will receive manual based sessions for sleeping disorders. The group meets once a week during six weeks according to following program:
  Session 1 - introduction, self-help concept Session 2 - biology of sleep, sleep restriction, Session 3 - stimulus control Session 4 - visualization as relaxation, Session 5 - how to deal with negative and automatic thoughts, Session 6 - how to solve problems, planning for the future
  Arms: Cognitive behavioral therapy (CBT)

SUMMARY:
"Auricular acupuncture and cognitive behavioral therapy in the context of insomnia and low dose dependence of benzodiazepine-like drugs and other sleep medicine with addiction risk"

INTRODUCTION: Insomnia is a common health problem in Sweden, which increases with age and is more prevalent among women.

It is defined by unsatisfied sleep quality during more than a month's time. The main symptoms are difficulties falling- and/or maintaining sleep, involuntary awakenings during the night of early morning, day time sleepiness and decreased will for day time activity due to sleepiness. Insomnia is ranked to be the fifth most common cause of prescription of medicine at the outpatient clinics in general health care in Sweden. In 2008 a prevalence study was initiated in Sweden by the Swedish Council on Health Technology Assessment (SBU). The study showed that 24% of the Swedish population suffered from sleep disorders. Sleeping disorders can go on for many years and can therefore entail significant personal suffering.

Usually sleep medicine combined with general sleeping advices is the first-hand treatment for insomnia. However, according to SBU, first treatment should be non-pharmacological, for instance cognitive behavioral therapy (CBT). Despite this recommendation the prescribing of sleep medicine is still high.

There are studies that suggest auricular acupuncture (AA) to be an effective method to treat insomnia. However more evidence is needed to draw firm conclusions.

AIM: The aim of the study is to investigate if AA is as effective as CBT to treat insomnia for patients who have stopped using benzodiazepine-like sleep medicine.

METHOD: This is a randomized controlled study (RTC) including patients suffering from insomnia, with a low dose dependence of benzodiazepine-like drugs. The patients will be recruited from primary care and from an out-patient clinic specialized in sleeping disorders and also by add in the local news paper. The respondents will be randomized to one of two groups; group I will receive AA twice a week for 4 weeks; group II will receive CBT once a week for six weeks. After three months there will be a long-time follow up in order to investigate a potential long-term effect.

DETAILED DESCRIPTION:
INTRODUCTION During the 1960s benzodiazepines were introduced in the health care. The benzodiazepines replaced the barbiturates because of their low toxicity and their anxiety reducing effect. During the 1990s the benzodiazepines were replaced with benzodiazepine-like drugs to treat insomnia. In Swedish health care two out of three recipes of hypnotics are prescribed to women, more than 50% of these are prescribed to persons of age > 65. To minimize the risk of drug tolerance a short time use of benzodiazepine-like drugs are recommended, and only after careful consideration from the prescriber. The risk of developing addiction is increased for people with prior substance dependence issues, people suffering from other psychiatric of mental health issues and for people with a high-dose intake.

Insomnia is a common symptom for people who suffer from substance dependence, especially when the intake has ended. During this time, the withdrawal phase, risk for relapse is high. The protracted withdrawal phase can go on for 6-12 months. General symptoms during this time, except insomnia, are sensitivity to stress, emotional over- and under reactions and memory dysfunctions.

Insomnia and drug dependence Insomnia is a common health problem in Sweden, which increases with age and is more prevalent among women.

Insomnia is defined by unsatisfied sleep quality during more than a month's time. The main symptoms are difficulties falling- and/or maintaining sleep, involuntary awakenings during the night of early morning, day time sleepiness and decreased will for day time activity due to sleepiness.

Sleep quality is, according to the National Board of Health and Welfare, a measurement of life quality among the population. Insomnia is ranked to be the fifth most common cause of prescription of medicine at the outpatient clinics in general health care in Sweden. In 2008 a prevalence study was initiated in Sweden by the Swedish Council on Health Technology Assessment (SBU). The study showed that 24% of the Swedish population suffered from sleep disorders. Sleeping disorders can go on for many years and can therefore entail significant personal suffering.

Sleeping disorders is treated by identifying the root cause, which can for instance be circadian disruption, life style factors, physiological- and psychological disease or side effects from drug treatment. Usually sleep medicine combined with general sleeping advices is the first-hand treatment. However, according to SBU, first treatment should be non-pharmacological, for instance cognitive behavioral therapy (CBT). Despite this recommendation the prescribing of sleep medicine is still high.

Acupuncture Acupuncture is a complementary (non-pharmacological) treatment method with roots in Traditional Chinese Medicine (TCM). The method is used as a stand alone treatment or as a complementary treatment for several types of health problems, for example to relieve pain, as a support for assisted conception, in chronic asthma treatment, and in schizophrenia treatment. In Sweden it is a part of the integrative methods within the health care, mostly used to relive pain or as assisting treatment during child birth.

Auricular acupuncture (AA) A later branch of traditional acupuncture is auricular acupuncture. The auricular method can be used to treat a wide variety of conditions, among others depression and insomnia. Auricular acupuncture involves inserting thin solid needles at selected points of the outer ear. In the late 1970's a specific auricular acupuncture protocol was developed to alleviate acute- and protracted withdrawal symptoms from opiate dependence and/or while adjusting methadone dose, now defined as the NADA (National Acupuncture Detoxification Association)-protocol. In Sweden, the NADA protocol is used as a complement to ordinary treatment in psychiatric care and in the context of protracted withdrawal symptoms from usage of alcohol and benzodiazepines.

Cognitive Behavior Therapy (CBT) CBT is a collective term for theories and techniques based upon learning psychology principles. By using different techniques the therapist and the patient can work with both situational- and/or long-term behavioral problems, for instance sleeping disorders. Treating sleeping disorders with CBT can be done through manual based group sessions.

Actigraphy Actigraphy is a way to measure sleep, circadian rhythm and activity and the measurement is done by the wrist of the persons' non-dominant hand. The device, which is similar to a wrist watch, registers the carriers' activity pattern during the days and nights. It can distinguish between sleep and activity and the information is processed through computer.

Present status report The Cochrane Library present a meta analyse in which auricular acupuncture has been used to treat insomnia. According to the result both auricular acupuncture and acupressure can improve sleep quality compared to placebo. However no firm conclusions could be made because of the low methodological quality of the studies. In order to draw conclusions, further research in the field is needed. In Sweden further research regarding complementary treatment methods to treat insomnia are requested by the SBU. Since insomnia is an increasing health problem in Sweden, the SBU also emphasize the importance of developing non-pharmacological treatment methods for insomnia in order to decrease substance dependence.

AIM The aim of the study is to investigate if AA is as effective as CBT to treat insomnia for patients who have stopped using benzodiazepine-like sleep medicine.

Question formulations

1. How are the sleep pattern, day/night activity and subjective sleep quality affected by AA treatment, alternative CBT, among women and men with a substance dependence of a prescribed therapeutic dose of benzodiazepine-like sleeping drugs?
2. Does the subjective quality of life change among women and men with a substance dependence of a prescribed therapeutic dose of benzodiazepine-like sleeping drugs, after treatment with AA or CBT, and if so, are there gender differences?
3. Is there a remaining effect of treatment 3 months after intervention has ended?

METHOD This is a randomized controlled study (RTC) including patients suffering from insomnia, with a low dose dependence of benzodiazepine-like drugs. The patients will be recruited from primary care and from out-patient clinic specialized in sleeping disorders and also by add in the local news paper. Once respondents are included in the study baseline will be measured regarding prevalence of insomnia, anxiety and depression. Other measurements are subjective perception of sleep- and life quality. Actigraphy will be used to monitor the respondents' activity pattern 24 hours a day for 7 days. The respondents will also use sleeping diaries. After baseline measurements the respondents end their sleeping medicine treatment. They will be randomized to one out of two groups.

Group I will receive AA and group II will receive CBT.

Inclusion criteria's: men and women (n=40) 18-75 years old with (i) primary or secondary insomnia who have been treated every day for over six months with benzodiazepine-like drugs and developed a low dose drug dependence, and (ii) people suffering from insomnia who use benzodiazepine-like drugs ≥ three nights a week with no effect.

Exclusion criteria's: high dose drug dependence, generalized anxiety disorder (GAD), patients diagnosed with diagnosed psychotic disorders, personality disorders or serious somatic illness, alcohol dependence/abuse, anti psychotic medications, pain reliving treatment with methadone- or methadone like drugs, new onset depression, patients who have initiated or changed their anti-depressant-, anxiolytic- or pregabalin medication during the last six months, pregnancy.

Questionnaires:

Hospital Anxiety Depression scale (HADs) prevalence of anxiety and depression, Insomnia Severity Index (ISI) prevalence of insomnia and effect of treatment, Minimal Insomnia Symptom Scale (MISS) prevalence of insomnia and effect of treatment, Functional Outcome of Sleep Questionnaire (FOSQ) measure consequences of sleepiness, Ep-worth Sleepless scale (ESS) measure sleepiness during day time, Form SF-12 measure quality of life, Dysfunctional Belief About Sleep (DBAS-16) measurement of subjective perception of sleep/lack of sleep.

After three months there will be a long-time follow up with actigraphy monitoring, sleeping diary and all questionnaires, in order to investigate a potential long-term effect.

Importance of the project Despite lack of scientific evidence AA is used nationally and internationally to treat conditions of substance dependence and of insomnia. According to patients and medical staff AA is perceived as at treatment method with positive and sometimes remaining results in the conditions mentioned above. The benefits of AA are the lack of severe side effects and the method is easy for the medical staff to learn how to perform. It is also a low cost method. Previous Swedish study within the substance dependence care showed that patients who had received AA treatment during protracted withdrawal, experienced that their subjective perceived sleep quality was improved. Since sleeping problems in many cases can lead to relapse in substance abuse, AA may be an eligible, non-pharmacological option for patients with high-risk profiles of developing substance dependence from sleeping drugs. If AA can contribute to a decreased risk of relapse in substance dependence and increase quality of life, the treatment can be of importance not only for individuals, but also in a health economical perspective and for society in general. The result of this project may contribute to strengthen the evidence for using AA to treat insomnia. From a public health perspective the method could, because of its lack of side effects, be an alternative treatment method that could be provided from the public health care.

ELIGIBILITY:
Inclusion Criteria:

* men and women (n=40)
* 18-75 years old with: (i) primary or secondary insomnia who have been treated every day for over six months with benzodiazepine-like drugs and developed a low dose drug dependence, and (ii) people suffering from insomnia who use benzodiazepine-like drugs ≥ three nights a week with no effect.

Exclusion Criteria:

* high dose drug dependence,
* generalized anxiety disorder (GAD),
* patients diagnosed with diagnosed psychotic disorders,
* personality disorders or serious somatic illness,
* alcohol dependence/abuse,
* anti psychotic medications,
* pain reliving treatment with methadone- or methadone like drugs,
* new onset depression,
* patients who have initiated or changed their anti-depressant,anxiolytic or pregabalin medication during the last six months,
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Insomnia | five months
  Outcome will be measured by:
  i)actigraphy ii)evaluated questionary forms: Insomnia Severity Index (ISI) Hospital Anxiety Depression scale (HAD) Minimal Insomnia Symptom Scale (MISS) Ep-worth Sleepless scale (ESS) Dysfunctional Belief About Sleep (DBAS-16) Functional Outcome of Sleep Questionaire (FOSQ)

SECONDARY OUTCOMES:
Quality of life | five months
  Quality of life will be measured by using "Form SF-12".

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Markström, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Bergdahl L, Broman JE, Berman AH, Haglund K, von Knorring L, Markstrom A. Auricular Acupuncture and Cognitive Behavioural Therapy for Insomnia: A Randomised Controlled Study. Sleep Disord. 2016;2016:7057282. doi: 10.1155/2016/7057282. Epub 2016 May 8. PMID 27242930